CLINICAL TRIAL: NCT01729767
Title: Assessment of Acyclovir Efficacy Versus Placebo in Controlling Vertigo Attacks of Patients With Meniere's Disease Visited in Amiralam Hospital
Brief Title: Efficacy of Antiviral Medications in Controlling Vertigo Attacks of Patients With Meniere's Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 88-03-48-9453
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Meniere's Disease
MeSH Terms: conditions — Meniere Disease | interventions — Acyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Acyclovir (Experimental): Acyclovir 400 mg tablets by mouth 5 times a day for the first month, 3 times a day for next 10 days, and 2 times a day for the last 10 days.
  Interventions: Drug: Acyclovir
- Placebo (Placebo Comparator): Placebo tablets by mouth 5 times a day for the first month, 3 times a day for next 10 days, and 2 times a day for the last 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acyclovir — Patients who were randomly allocated to the Acyclovir group besides sticking with low salt diet will take the Acyclovir 400 mg pills for 10 days 5 times a day, then 3 times a day for next 10 days, and 2 times a day for the last 10 days. Patients would receive the medication in 2 sessions, first in the beginning of the study and the rest after 10 days. This way it would boost their compliance, and physicians would be aware of possible complications. Patients will report changes in their symptoms 10 days after initiating the drug and in 1, 3, and 6 month intervals. All changes in frequency and duration of vertigo attacks are recorded, and their tinnitus and aural fullness is recorded in a 0(with no symptom) to 4 (very severe) scale.
  Other Names: Zovirax
  Arms: Acyclovir
Drug: Placebo — Participants who are randomly placed in placebo group, besides sticking with low salt diet will take the placebo (inert ingredient) for 10 days 5 times a day, then 3 times a day for next 10 days, and 2 times a day for the last 10 days. Patients would receive the medication in 2 sessions, first in the beginning of the study and the rest after 10 days. This way it would boost their compliance, and physicians would be aware of possible complications. Patients will report changes in their symptoms 10 days after initiating the drug and in 1, 3, and 6 month intervals. All changes in frequency and duration of vertigo attacks are recorded, and tinnitus and aural fullness is recorded in a 0(with no symptom) to 4 (very severe) scale.
  Other Names: sugar pills, manufactured to mimic the Acyclovir 400 mg tablets.
  Arms: Placebo

SUMMARY:
Meniere's disease is a chronic illness that affects a substantial number of patients every year worldwide. The disease is characterized by intermittent episodes of vertigo lasting from minutes to hours, with fluctuating sensorineural hearing loss, tinnitus, and aural pressure. It has recently been suggested that viral etiologies specially Herpes virus might be the underlying reason. The investigators study is a randomized, double- blinded placebo-controlled clinical trial in Amiralam Hospital. In this study the primary objective is to assess efficacy of Acyclovir in control of symptoms in patients with Meniere's disease specially their vertigo attacks. Inclusion criteria would be patient's willingness to participate in the study and follow ups, being 18 years old or older, having at least 2 vertigos per month each at least 20 min, interfering with function, and not on medication for Meniere's disease for at least 3 months before the trial. They should not have any history of allergy to Acyclovir, renal insufficiency or Creatinine above 1.5 mg/dl, hepatic enzymes more than three times normal, serious uncontrolled illness, be pregnant or nursing or have previous surgeries on Endolymphatic Sac. Participants will be randomly placed in 2 different arms getting either Acyclovir 400 mg or placebo (inert ingredient). They will take the medication for 10 days 5 times a day, then 3 times a day for next 10 days, and 2 times a day for the last 10 days. Patients will report changes in their symptoms 10 days after initiating the drug and in 1, 3, 6 month intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' willingness to participate in the study
2. Willingness to participate in follow ups
3. Age of 18 or older
4. Having at least 2 vertigos per month each lasting for at least 20 min, severely interfering with function
5. Not on medication for at least 3 months before starting the trial

Exclusion Criteria:

1. History of Allergy to Acyclovir or the drugs in the same category
2. Renal insufficiency or having Creatinine more than 1.5 mg/dl
3. Hepatic enzymes more than 3 times normal
4. Hematocrit less than 30%
5. Thrombocytopenia
6. Having a serious uncontrolled illness
7. Pregnant or nursing ladies
8. Using Probenecid
9. Previous surgeries on Endolymphatic Sac.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Vertigo | Change from baseline after 3 months

SECONDARY OUTCOMES:
Hearing Loss | Change from baseline after 3 months
  Method of measurement would be Audiometry and also subjective evaluation
Aural Fullness | Change from baseline after 3 months
  Method of measurement would be subjective evaluation in a 0 (with no symptom) to 4 (very severe) scale
Tinnitus | Change from baseline in 3 months
  Method of measurement would be subjective evaluation in a 0 (with no symptom) to 4 (very severe) scale

CONTACTS AND LOCATIONS:
Locations (1):
- Amiralam Hospital, Tehran, Iran